CLINICAL TRIAL: NCT02739373
Title: Randomized, Double-Blinded, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Pharmacodynamics of BMS-986189 in Healthy Subjects
Brief Title: Pharmacokinetics, Safety, Tolerability and Pharmacodynamics of BMS-986189 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AI006-003
Record Dates: First submitted 2016-04-08; First posted 2016-04-15 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-986189 (Experimental): Specified Dose on Specified Day
  Interventions: Drug: BMS-986189
- Placebo (Placebo Comparator): Specified Dose on Specified Day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986189
  Arms: BMS-986189
Other: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to measure the amount of study drug (BMS-986189) in the blood and urine and to see if BMS-986189 is safe and well-tolerated in healthy people after a single dose.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy, males and females, 18 to 55 years of age, inclusive
* Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, inclusive
* Women of childbearing potential (WOCBP) must have negative serum pregnancy test (performed for all females; minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to start of study drug

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of diabetes mellitus, severe hypertriglyceridemia, acute or chronic pancreatitis, pancreatic exocrine disorder
* History of autoimmune disease
* Any known skin condition that would affect subcutaneous dosing
* Positive blood screen for hepatitis C antibody (HCV Ab), hepatitis B surface antigen (HBsAg), or HIV -1 and HIV -2 antibody

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Day 1 to Day 30
Time of maximum observed concentration (Tmax) | Day 1 to Day 30
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(O-T)) | Day 1 to Day 30
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Day 1 to Day 30
Half Life (T-HALF) | Day 1 to Day 30
Total Body Clearance (CLT/F) | Day 1 to Day 30
Apparent volume of distribution at steady state (Vss/F) | Day 1 to Day 30
Deaths leading to discontinuation | Day 1 to Day 30
Adverse events (AEs) leading to discontinuation | Day 1 to Day 30
Serious adverse events (SAEs) leading to discontinuation | Day 1 to Day 30
Lab abnormalities leading to discontinuation | Day 1 to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit, Inc., Evansville, Indiana, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx